CLINICAL TRIAL: NCT01011413
Title: A Randomised, Double-blind, Placebo-controlled, Trial to Compare the Safety and Efficacy of Reduced Dose Versus Standard Dose EFV Plus Two Nucleotides (N(t)RTI) in Antiretroviral-naïve HIV-infected Adults Over 96 Weeks
Brief Title: Safety and Efficacy of Reduced Versus Standard Dose Efavirenz (EFV) Plus Two Nucleotides in Antiretroviral-naïve Adults.
Acronym: ENCORE1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCHECR-ENCORE1
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: HIV Infections
Keywords: HIV; Antiretroviral Therapy (ART); Efavirenz (EFV); Dose reduction
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 600 milligram (mg) Efavirenz (Active Comparator): Eligible patients will be centrally randomised to receive tenofovir (TDF) (300mg qd)/emtricitabine (FTC) (200mg qd) + EFV (600mg qd; 3 x 200mg qd)
  Interventions: Drug: Efavirenz 600mg
- 400mg Efavirenz (Experimental): Eligible patients will be centrally randomised to receive TDF (300mg qd)/FTC (200mg qd) + EFV (400mg qd; 2 x 200mg + 1 x 200mg placebo qd).
  Interventions: Drug: Efavirenz 400mg

INTERVENTIONS:
Drug: Efavirenz 600mg — 3 x EFV 200 milligram (mg) tablets once daily
  Other Names: Matrix EFV 200mg tablets
  Arms: 600 milligram (mg) Efavirenz
Drug: Efavirenz 400mg — 2 x EFV 200 milligram (mg) tablets plus 1x matched EFV placebo tablet once daily
  Other Names: Matrix EFV 200mg tablets; Matrix EFV 200mg matched placebo tablets.
  Arms: 400mg Efavirenz

SUMMARY:
Clinical data suggests that the standard dose of the anti-HIV medication, efavirenz (EFV), could be reduced without compromising its effectiveness. Lower drug doses could have fewer side effects and would make EFV more affordable. The purpose of this study is to compare the safety and effectiveness, over 96 weeks, of standard (600mg) versus reduced dose (400mg) EFV in controlling HIV as part of initial combination antiretroviral therapy.

DETAILED DESCRIPTION:
In this international, multicenter trial, 630 HIV infected patients who have not received any previous treatment for their HIV-infection will be enrolled. Participants will be randomized equally (1:1) to receive Truvada (tenofovir and emtricitabine) with either the standard or reduced dose of EFV. Neither the study doctor nor the participant will know which treatment the participant is receiving. Physical examinations, laboratory analyses and questionnaires will be performed at the 11 study visits at screening, baseline (Week 0), Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96. The primary aim of this study is to compare between treatment groups the proportion of patients with undetectable HIV viral load (HIV RNA < 200 copies/mL) after 48 weeks. Information on immune function, drug adherence, resistance to antiretrovirals, quality of life, mental state and HIV-related conditions will also be collected. Blood samples will be collected for future testing. Interim analyses will be performed when the first 125 participants in each treatment group reach week 24 and when all participants reach week 24. These interim analyses will provide an early check that the reduced dose of EFV suppresses HIV infection as effectively as the standard dose of EFV. A follow-up analysis will be performed when all participants reach week 96.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive by licensed diagnostic test
* aged >16 years of age (or minimum age as determined by local regulations or as legal requirements dictate)
* 50 < cluster of differentiation (CD)4 <500 cells/µL
* No prior AIDS-defining illness, using the Center for Diseases Control 1993 Case Definition (except pulmonary tuberculosis)
* HIV RNA ≥1000 copies/mL
* no prior exposure to antiretroviral therapy (ART) (including short course ART for preventing MTCT)
* calculated creatinine clearance (CLCr) more than or equal to 50 mL/min (Cockcroft-Gault formula)
* provision of written informed consent.

Exclusion Criteria:

* the following laboratory values:

  * absolute neutrophil count (ANC) <500 cells/μL
  * hemoglobin <7.0 g/dL
  * platelet count <50,000 cells/μL
  * alanine aminotransferase and/or aspartate aminotransferase >5 x upper limit of normal
* pregnant women or nursing mothers
* active opportunistic or malignant disease not under adequate control
* use of immunomodulators within 30 days prior to screening
* use of any prohibited medications
* current alcohol or illicit substance use that might adversely affect study participation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Cooper, Professor, Principal Investigator — Kirby Institute
Locations (1):
- St Vincent's Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Result] ENCORE1 Study Group. Efficacy of 400 mg efavirenz versus standard 600 mg dose in HIV-infected, antiretroviral-naive adults (ENCORE1): a randomised, double-blind, placebo-controlled, non-inferiority trial. Lancet. 2014 Apr 26;383(9927):1474-1482. doi: 10.1016/S0140-6736(13)62187-X. Epub 2014 Feb 10. PMID 24522178
- [Result] ENCORE1 Study Group; Carey D, Puls R, Amin J, Losso M, Phanupak P, Foulkes S, Mohapi L, Crabtree-Ramirez B, Jessen H, Kumar S, Winston A, Lee MP, Belloso W, Cooper DA, Emery S. Efficacy and safety of efavirenz 400 mg daily versus 600 mg daily: 96-week data from the randomised, double-blind, placebo-controlled, non-inferiority ENCORE1 study. Lancet Infect Dis. 2015 Jul;15(7):793-802. doi: 10.1016/S1473-3099(15)70060-5. Epub 2015 Apr 12. PMID 25877963
- [Derived] Winston A, Amin J, Clarke A, Else L, Amara A, Owen A, Barber T, Jessen H, Avihingsanon A, Chetchotisakd P, Khoo S, Cooper DA, Emery S, Puls R; ENCORE Cerebrospinal Fluid (CSF) Substudy Team; ENCORE Cerebrospinal Fluid CSF Substudy Team. Cerebrospinal fluid exposure of efavirenz and its major metabolites when dosed at 400 mg and 600 mg once daily: a randomized controlled trial. Clin Infect Dis. 2015 Apr 1;60(7):1026-32. doi: 10.1093/cid/ciu976. Epub 2014 Dec 11. PMID 25501988
- See also: Kirby Institute (formerly National Centre for HIV Epidemiology and Clinical Research) — https://kirby.unsw.edu.au

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 clinical centres (primary and tertiary care facilities) in 13 countries on 5 continents screened a total of 768 patents who had provided informed consent between Aug 4, 2011 and March 19, 2012.
Pre-assignment Details: 768 screened:132 did not satisfy eligibility: 2 prior AIDS-defining illness; 3 previous antiretroviral therapy; 15 HIV RNA out of range; 44 cluster of differentiation (CD)4 count out of range; 13 lab values out of range; 2 pregnant; 9 intercurrent illness; 2 illicit substance use; 30 exceeded screen time; 4 clinician exclusion; 9 withdrew consent.
Groups:
- 600mg Efavirenz: Eligible patients will be centrally randomised to receive tenofovir (TDF) (300mg qd)/emtricitabine (FTC) (200mg qd) + EFV (600mg qd; 3 x 200mg qd)
  Efavirenz: 3 x EFV 200mg tablets once daily
- 400mg Efavirenz: Eligible patients will be centrally randomised to receive TDF (300mg qd)/FTC (200mg qd) + EFV (400mg qd; 2 x 200mg + 1 x 200mg placebo qd).
  Efavirenz: 2 x EFV 200mg tablets plus 1x matched EFV placebo tablet once daily
Period: Overall Study
Arm/Group | 600mg Efavirenz | 400mg Efavirenz
Started | 312 (312 randomised) | 324 (324 randomised)
Did Not Start Study Drug | 3 | 3
In Modified ITT | 309 | 321
Died Before Week 48 | 3 | 2
Lost to Follow up Before w48 | 3 | 4
Withdrew Consent Before w48 | 3 | 3
Attended w48 Visit | 295 | 311
Died Between Week 48 and 96 | 2 | 3
Withdrew Consent Between Week 48 and 96 | 2 | 6
Lost to Follow-up Between Week 48 and 96 | 10 | 4
Completed | 286 | 299
Not Completed | 26 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 600mg Efavirenz | 400mg Efavirenz | Total
Number analyzed (Participants) | 309 | 321 | 630
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (10.0) | 36.1 (10.0) | 36.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 100 | 203
  Male | 206 | 221 | 427
Race/Ethnicity, Customized [Number; unit: participants]
  African | 116 | 118 | 234
  Asian | 103 | 106 | 209
  White | 90 | 97 | 187
HIV transmission risk [Number; unit: participants]
  heterosexual | 156 | 156 | 312
  homo/bisexual | 134 | 138 | 272
  injecting drug user/not known | 19 | 27 | 46
CDC HIV infection clinical category [Number; unit: participants] — As assessed by the Centres for Disease Control and Prevention (CDC) 1993 Revised Classification System for HIV Infection for Adolescents and Adults. Published in Morbidity and Mortality Weekly Report December 18, 1992 / 41(RR-17). Clinical category of HIV infection was assigned by the clinician based on the clinical conditions that define each of the three categories. Category A is the best, followed by category B and lastly category C.
  participants
    category A | 265 | 264 | 529
    category B | 33 | 46 | 79
    category C | 11 | 11 | 22
Median plasma HIV RNA [Median (Inter-Quartile Range); unit: log10 copies per mL] | 4.73 [3.83 to 5.63] | 4.76 [3.92 to 5.60] | 4.75 [3.87 to 5.63]
Mean nadir cluster of differentiation (CD)4+ cell count [Mean (Standard Deviation); unit: cells per mm3] | 252 (90) | 248 (88) | 250 (89)
Hep B Sag +ve [Number; unit: participants] — number of participants surface antigen positive
  participants | 12 | 15 | 27
Hep C ab +ve [Number; unit: participants] — number of participants antibody positive
  participants | 3 | 5 | 8
Mean creatinine clearance (mL/min) [Mean (Standard Deviation); unit: mL per min] | 120 (32.4) | 117.4 (29.7) | 118.7 (31.0)
Mean total chol (mmol/L) [Mean (Standard Deviation); unit: mmol per Litre] | 4.15 (0.93) | 4.24 (0.95) | 4.20 (0.94)
Mean HDL chol (mmol/L) [Mean (Standard Deviation); unit: mmol per Litre] | 1.03 (0.31) | 1.04 (0.32) | 1.03 (0.32)
Mean LDL chol (mmol/L) [Mean (Standard Deviation); unit: mmol per Litre] | 2.47 (0.84) | 2.54 (0.93) | 2.51 (0.88)
Mean triglycerides (mmol/L) [Mean (Standard Deviation); unit: mmol per Litre] | 1.24 (0.69) | 1.25 (0.72) | 1.25 (0.70)
Insulin (mU/L) [Mean (Standard Deviation); unit: mU per Litre] | 8.28 (9.70) | 8.26 (12.9) | 8.27 (11.4)
Glucose (mmol/L) [Mean (Standard Deviation); unit: mmol per Litre] | 4.84 (1.78) | 4.66 (0.98) | 4.75 (1.43)
Current smoker [Number; unit: participants] | 87 | 82 | 169
Mean BMI (kg/m^2) [Mean (Standard Deviation); unit: kg per m2] | 24.3 (5.2) | 24.0 (4.7) | 24.2 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HIV-1 RNA <200 Copies/mL 48 Weeks After Randomisation
Description: Percentage of participants in each of the treatment arms with centrally quantified plasma HIV-1 RNA viral load <200 copies/mL 48 weeks after randomisation.
Time Frame: 48 weeks
Population: modified intention to treat including all randomised patients who took at least one dose of study medication AND attended at least one follow-up visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 600mg Efavirenz: Efavirenz: 3 x EFV 200mg tablets once daily plus tenofovir/emtricitabine 300 mg/200 mg
- 400mg Efavirenz: Efavirenz: 2 x EFV 200mg tablets plus 1x matched EFV placebo tablet once daily plus tenofovir/emtricitabine 300 mg/200 mg
Arm/Group | 600mg Efavirenz | 400mg Efavirenz
Number analyzed (Participants) | 309 | 321
percentage of participants | 92.2 [89.2 to 95.2] | 94.1 [91.5 to 96.7]
Statistical Analysis 1: Comparison: 600mg Efavirenz vs 400mg Efavirenz; Sample size calculation assumes 85% of participants randomised to 600mg EFV arm will have plasma HIV RNA <200 copies/ml at 48 weeks. Assuming no difference between randomised treatments in proportion with plasma HIV RNA <200 copies/mL, to have 90% power to demonstrate non-inferiority in the intention to treat (ITT) analysis using a 10% non-inferiority margin will require 286 participants per arm, making a total of 572 participants. Power for modified ITT analysis was 93%; Test type: Non-Inferiority — Only the primary endpoint is assessed in terms of non-inferiority. All other comparisons are tests for superiority and are considered statistically significant at a two-sided alpha=0.05. Non-inferiority of EFV 400 mg was defined as the lower 95% confidence interval (CI) of the difference between groups in the proportion of viral load below 200 copies/mL at week 48 lying above -10%; p = 0.05, Pearson's chi-squared — No adjustments were made for multiple comparisons; Pearson's chi-squared or Fisher's exact test derived p value was used
Statistical Analysis 2: Comparison: 600mg Efavirenz vs 400mg Efavirenz; To ensure the per protocol (PP) analysis has 90% power to demonstrate non-inferiority, the sample size was inflated for patients who switch treatment for toxicity. This is estimated to be no more than 10% randomised patients. To ensure 90% power to demonstrate non-inferiority in the ITT and PP analyses, a total of 630 (315 per arm) patients will be randomised giving 93% power for the ITT analysis. Null hypothesis: no statistically significant difference between the 600mg and 400mg EFV regimens; Test type: Non-Inferiority — Non-inferiority will be defined as the lower 95% confidence limit of the difference in percentages of patients with undetectable viral load lying above -10% (i.e. a non-inferiority margin of 10%); p = 0.05, Chi-squared — No adjustment for multiple comparisons

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <400 Copies/mL and <50 Copies/mL at 48 and 96 Weeks After Randomisation
Description: Percentage of participants in each of the two treatment arms with plasma HIV-1 RNA <400 copies/mL and <50 copies/mL at 48 and 96 weeks after randomisation
Time Frame: Baseline and 2 years
Population: Modified ITT including all randomised participants who took at least one dose of study medication and attended at least one follow-up visit
Measure: Number; unit: participants
Groups:
- 600 mg Efavirenz: EFV 600 mg plus tenofovir 300 mg and emtricitabine 200 mg daily
- Efavirenz 400 mg: EFV 400 mg plus tenofovir 300 mg and emtricitabine 200 mg daily
Arm/Group | 600 mg Efavirenz | Efavirenz 400 mg
Number analyzed (Participants) | 309 | 321
participants
  HIV-1 RNA <50cp/mL | 268 | 277
  HIV-1 RNA <400cp/mL | 280 | 291
Statistical Analysis 1: Comparison: 600 mg Efavirenz vs Efavirenz 400 mg; Test type: Superiority or Other; p = 0.05, Chi-squared — P-value not adjusted for multiple comparisons; difference between proportions = 0.05

3. Secondary Outcome: Mean Change From Baseline in CD4+ T-cell Count
Description: Mean change from baseline to week 96 in CD4+ T-cell count/mm3 between the two treatment arms
Time Frame: Baseline and 2 years
Population: modified ITT (all participants who received at least one dose of study treatment and attended at least one follow up visit, irrespective of treatment received)
Measure: Mean (95% Confidence Interval); unit: cells per mm3
Groups:
- 600mg Efavirenz: Efavirenz 600mg: 3 x EFV 200 mg tablets once daily plus tenofovir/emtricitabine 300 mg /200 mg
- 400mg Efavirenz: Efavirenz 400 MG: 2 x EFV 200 milligram (mg) tablets plus 1x matched EFV placebo tablet once daily plus tenofovir/emtricitabine 300 mg/200 mg
Arm/Group | 600mg Efavirenz | 400mg Efavirenz
Number analyzed (Participants) | 309 | 321
cells per mm3 | 209 [194 to 226] | 235 [218 to 252]

4. Secondary Outcome: Clinical Endpoints: Opportunistic Disease or Death, and Serious Non-AIDS-defining Events and Non-AIDS-related Mortality
Description: Number of participants in each randomised arm diagnosed with a serious non-AIDS defining event, who die from an AIDS-defining event, who die from a non-AIDS-defining event
Time Frame: up to 2 years
Population: modified ITT population
Measure: Count of Participants; unit: Participants
Groups:
- 600mg Efavirenz: Efavirenz 600mg: 3 x EFV 200 mg tablets once daily plus tenofovir/emtricitabine 300 mg/200 mg
- 400mg Efavirenz: Efavirenz 400 MG: 2 x EFV 200mg tablets plus 1x matched EFV placebo tablet once daily plus tenofovir/emtricitabine 300 mg/200 mg
Arm/Group | 600mg Efavirenz | 400mg Efavirenz
Number analyzed (Participants) | 309 | 321
Participants
  AIDS events | 7 | 14
  AIDS event deaths | 2 | 0
  non-AIDS deaths | 5 | 3
  serious non-AIDS events | 3 | 3
  No disease/death | 292 | 301

5. Secondary Outcome: Change From Baseline in Metabolic Endpoints
Description: Change from baseline to week 96 in fasted total cholesterol, high density cholesterol and low density cholesterol, and glucose between randomised treatment arms
Time Frame: Baseline and 2 years
Population: Available data analysis
Measure: Mean (95% Confidence Interval); unit: mmol per Litre
Groups:
- 600mg Efavirenz: Efavirenz 600mg: 3 x EFV 200mg once daily plus tenofovir/emtricitabine 300 mg/200 mg tablets once daily
Arm/Group | 600mg Efavirenz | 400mg Efavirenz
Number analyzed (Participants) | 309 | 321
mmol per Litre
  Total cholesterol mmol/L: number analyzed (Participants) | 279 | 292
  Total cholesterol mmol/L | 0.62 [0.53 to 0.71] | 0.54 [0.44 to 0.63]
  HDL mmol/L: number analyzed (Participants) | 273 | 286
  HDL mmol/L | 0.35 [0.31 to 0.40] | 0.30 [0.26 to 0.34]
  LDL mmol/L: number analyzed (Participants) | 271 | 283
  LDL mmol/L | 0.21 [0.13 to 0.29] | 0.16 [0.09 to 0.23]
  Blood glucose mmol/L: number analyzed (Participants) | 281 | 293
  Blood glucose mmol/L | 0.24 [0.07 to 0.4] | 0.40 [0.30 to 0.50]

6. Secondary Outcome: Adherence: Median Scores of Self-reported Adherence to Randomised Study Medications
Description: AIDS Clinical Trials Group (ACTG) 7-day adherence questionnaire scores. Maximum value is all pills taken every day; minimum value is no pills taken per day. Higher scores indicate a better outcome.
Time Frame: 2 years
Population: Number of participants attending week 96 visit
Measure: Count of Participants; unit: Participants
Arm/Group | 600mg Efavirenz | 400mg Efavirenz
Number analyzed (Participants) | 280 | 292
Participants
  All pills taken | 256 | 271
  Most pills taken | 7 | 12
  About half pills taken | 1 | 1
  No pills taken | 16 | 8

7. Secondary Outcome: Change From Baseline in Fasted Insulin Levels
Description: Change from baseline to week 96 in fasted insulin levels
Time Frame: Baseline and 2 years
Population: Available data analysis
Measure: Mean (95% Confidence Interval); unit: mU per litre
Arm/Group | 600mg Efavirenz | 400mg Efavirenz
Number analyzed (Participants) | 309 | 321
mU per litre | -0.11 [-0.23 to 1.02] | 0.3 [-1.81 to 2.42]

8. Secondary Outcome: Change in Selected Serum Biochemical Parameters
Description: Change from baseline to week 96 in alanine aminotransferase, aspartate aminotransferase and alkaline phosphatase levels between randomised treatment arms
Time Frame: Baseline and 2 years
Population: Available data analysis
Measure: Mean (95% Confidence Interval); unit: Units per Litre
Arm/Group | 600 mg Efavirenz | Efavirenz 400 mg
Number analyzed (Participants) | 309 | 321
Units per Litre
  Alanine aminotransferase: number analyzed (Participants) | 285 | 298
  Alanine aminotransferase | 6.53 [1.04 to 12.02] | 0.64 [-3.52 to 4.79]
  Aspartate aminotransferase: number analyzed (Participants) | 283 | 297
  Aspartate aminotransferase | 1.71 [-1.69 to 5.10] | -1.23 [-3.67 to 1.21]
  Alkaline phosphatase: number analyzed (Participants) | 284 | 299
  Alkaline phosphatase | 26.75 [22.9 to 30.61] | 21.23 [17.4 to 25.05]

9. Secondary Outcome: Change From Baseline in Estimate Creatinine Clearance
Description: Change from baseline to week 96 in estimate creatinine clearance between randomised treatment arms
Time Frame: Baseline and 2 years
Population: Available data analysis
Measure: Mean (95% Confidence Interval); unit: millilitres per minute
Arm/Group | 600mg Efavirenz | 400mg Efavirenz
Number analyzed (Participants) | 309 | 321
millilitres per minute | -0.17 [-2.45 to 2.10] | 1.59 [-1.05 to 4.24]

10. Secondary Outcome: Steady-state Efavirenz Concentrations
Description: Steady-state efavirenz mid-dosing interval plasma concentrations
Time Frame: Week 4
Population: Available data analysis
Measure: Geometric Mean (90% Confidence Interval); unit: milligram per Litre
Arm/Group | 600mg Efavirenz | 400mg Efavirenz
Number analyzed (Participants) | 295 | 311
milligram per Litre | 2.85 [2.70 to 3.0] | 2.10 [2.01 to 2.20]

ADVERSE EVENTS:
Time Frame: 96 weeks. Analyses were modified intention-to-treat which included all randomised participants who received at least one dose of study drug and had at least one follow-up visit. Number of participants in the modified ITT analysis at week 96 are: 321 for EFV 400mg and 309 for EFV 600mg
Description: Adverse event analysis included all randomised participants who received at least one dose of study drug and had at least one follow-up visit. Number of participants in this modified ITT analysis at week 96 are: 321 for EFV 400mg and 309 for EFV 600mg
Arm/Group | 600mg Efavirenz | 400mg Efavirenz
All-Cause Mortality (participants affected / at risk) | 7/309 | 3/321
Serious Adverse Events (participants affected / at risk) | 25/309 | 23/321
Other Adverse Events (participants affected / at risk) | 273/309 | 286/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 600mg Efavirenz (N=309) | 400mg Efavirenz (N=321)
abscess (Infections and infestations) | 0 (0) | 1 (1)
bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
appendicitis (Infections and infestations) | 0 (0) | 1 (1)
bacterial diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 0 (0)
urosepsis (Infections and infestations) | 2 (2) | 0 (0)
dengue fever (Infections and infestations) | 1 (1) | 0 (0)
perianal abscess (Infections and infestations) | 1 (1) | 0 (0)
dizziness (Vascular disorders) | 0 (0) | 1 (1)
haemorrhoids (Vascular disorders) | 0 (0) | 1 (1)
gastrointestinal haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
cerebrovascular accident (Vascular disorders) | 1 (1) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
cerebral toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1)
disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
subdural haematoma (Vascular disorders) | 1 (1) | 0 (0)
testicular seminoma stage II (Reproductive system and breast disorders) | 1 (1) | 0 (0)
priapism (Reproductive system and breast disorders) | 0 (0) | 0 (0)
testicular injury (Reproductive system and breast disorders) | 0 (0) | 1 (1)
anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
pyrexia (General disorders) | 0 (0) | 2 (2)
lip oedema (Immune system disorders) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Immune system disorders) | 0 (0) | 1 (1)
nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
visual disturbance (Eye disorders) | 1 (1) | 0 (0)
hepatitis C (Hepatobiliary disorders) | 1 (1) | 0 (0)
skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0)
abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
rash macro-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
breast lump removal (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 600mg Efavirenz (N=309) | 400mg Efavirenz (N=321)
upper respiratory tract infection (Infections and infestations) | 36 (41) | 57 (68)
nasopharyngitis (Infections and infestations) | 18 (26) | 26 (30)
influenza (Infections and infestations) | 17 (22) | 18 (23)
gastroenteritis (Infections and infestations) | 13 (13) | 17 (19)
dizziness (Vascular disorders) | 107 (121) | 85 (96)
diarrhoea (Gastrointestinal disorders) | 36 (40) | 33 (38)
nausea (Gastrointestinal disorders) | 22 (24) | 14 (15)
rash (Skin and subcutaneous tissue disorders) | 41 (44) | 57 (65)
abnormal dreams (Psychiatric disorders) | 35 (35) | 28 (29)
insomnia (Psychiatric disorders) | 20 (21) | 20 (21)
headache (Nervous system disorders) | 34 (40) | 35 (44)
cough (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No